CLINICAL TRIAL: NCT07051447
Title: The Reducing Adverse Outcomes in Dialysis by Adjusting the pRescription for Dialysate Potassium Trial (RADAR-K): A Randomized, Controlled, Pilot Trial Comparing Usual Care to a Precision Approach to Dialysis Potassium Prescribing.
Brief Title: The Reducing Adverse Outcomes in Dialysis by Adjusting the pRescription for Dialysate Potassium Trial
Acronym: RADAR-K
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 24-01766
Record Dates: First submitted 2025-06-26; First posted 2025-07-04 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-06

CONDITIONS: End Stage Kidney Disease
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Dialysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Precision approach to K Prescription for HD (PKRxHD) (Experimental): Participants will receive a novel dialysate potassium (K) management strategy.
  Interventions: Other: PKRxHD; Procedure: Dialysis
- Usual Care (Active Comparator): Standard dialysis potassium prescribing.
  Interventions: Procedure: Dialysis

INTERVENTIONS:
Other: PKRxHD — The precision approach will incorporate point of care testing of blood potassium concentration prior to each dialysis session and adjustment of the dialysate K prescription with a blood-dialysate K gradient minimization strategy (PKRxHD).
  Arms: Precision approach to K Prescription for HD (PKRxHD)
Procedure: Dialysis — Standard of care dialysis.

SUMMARY:
This will be a randomized controlled pilot trial comparing usual care to a precision approach to dialysis potassium prescribing. The precision approach will incorporate point of care testing of blood potassium concentration prior to each dialysis session and adjustment of the dialysate K prescription with a blood-dialysate K gradient minimization strategy (PKRxHD).

ELIGIBILITY:
Inclusion Criteria:

* Undergoing in-center, 3x/weekly HD for treatment of end-stage kidney disease (ESKD) for at least 90 days
* Age at least 21 years
* Prescribed HD time up to 15 hours/ week

Exclusion Criteria:

* Incarcerated
* Life expectancy of 1 year or less
* Kidney transplant, transition to home dialysis, or transfer to non-participating HD unit anticipated within 6 months or less
* Cognitive condition that precludes consent
* Severe anemia (hemoglobin < 8.0 g/dL) within 30 days
* K concentration of 7.0 mEq/L or more within 60 days
* Pregnant women
* Women of childbearing potential actively trying to conceive unwilling to use contraception
* Participation in other interventional studies within 30 days prior to enrollment

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2029-02-01 (Estimated); Study Completion 2029-08-01 (Estimated)

PRIMARY OUTCOMES:
Intervention Adherence | Up to Week 24
  Measured as the proportion of hemodialysis (HD) treatments in the experimental arm completed per protocol with both pre-HD point of care testing and appropriate adjustment of the dialysate prescription.
Recruitment Feasibility | Baseline
  Measured as the proportion of eligible patients enrolled successfully.
Incidence Rate of Pre-HD Hyperkalemia | Baseline
  Hyperkalemia is defined as K≥ 6.4 mEq/L.
Post-HD Recovery Time | Up to Week 24
  Measured as the average time to recovery following each HD session.

SECONDARY OUTCOMES:
Incidence Rate of Post-HD Hyperkalemia Incidence Rate | Up to Week 24
  Hyperkalemia is defined as K≥ 6.4 mEq/L.
Incidence Rate of Moderate Hyperkalemia | Up to Week 24
  Hyperkalemia is defined as K≥ 3.0 mEq/L.
Incidence Rate of Peri-Dialytic Cramping | Up to Week 24
Incidence Rate of Intradialytic Hypotension | Up to Week 24
  Intradialytic hypotension will be defined as the proportion of HD sessions with intradialytic systolic blood pressure<90 mmHg, as this definition best captures associations with mortality according to current guidelines.

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset will be shared upon reasonable request beginning 9 to 36 months after publication or as required by a condition of awards or supporting agreements, provided the requesting investigator executes a data use agreement with NYU Langone Health. This instance of data sharing will also require separate IRB review as well as review from NYU Langone's Data Sharing Strategy Board (DSSB). Requests should be directed to: [contact information for PI or designee]. The protocol and statistical analysis plan will be posted on Clinicaltrials.gov only as required by federal regulation or supporting awards and agreements.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will be granted access upon reasonable request. Requests should be directed to David.Charytan@nyulangone.org. To gain access, data requestors will need to sign a data access agreement. This instance of data sharing will also require separate IRB review as well as review from NYU Langone's DSSB.